CLINICAL TRIAL: NCT04477304
Title: Application of Economics & Social Psychology to Improve Opioid Prescribing Safety Trial 1: Electronic Health Record Nudges
Brief Title: Application of Economics & Social Psychology to Improve Opioid Prescribing Safety Trial 1: EHR Nudges
Acronym: AESOPS-T1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Northwestern University (Other); AltaMed Health Services Corporation (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jason Doctor, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R33AG057395 (NIH); R33AG057395 (NIH)
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Opioid Abuse, Unspecified
Keywords: opioid use disorder; randomized control trial; behavioral economics; nudges
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention Arm (Experimental): Clinicians in clinics randomized to the intervention group will be prompted with an EHR nudge when the prescribing history for the patient falls into one of the following three categories: Opioid naïve, At-risk for long-term use, or Long-term opioid recipient. These EHR-based nudges include elements of accountable justification, defaults and precommitments. Clinicians will also receive web-based guideline education, consisting of an online educational module at the start of the study period. This will include educational clinical content related to the CDC guidelines, the Oregon Pain Guidance document, tapering training and other resources such as Substance Abuse and Mental Health Services Administration (SAMHSA) Medication-Assisted Treatment Physician Locator and the Naloxone Provider Guide.
  Interventions: Behavioral: Opioid Naive, OR; Behavioral: At-risk for long-term use, OR; Behavioral: Long-term opioid recipient
- Control (No Intervention): Clinicians in clinics randomized to the control group will receive web-based guideline education, consisting of an online educational module at the start of the study period. This will include educational clinical content related to the CDC guidelines, the Oregon Pain Guidance document, tapering training and other resources such as Substance Abuse and Mental Health Services Administration (SAMHSA) Medication-Assisted Treatment Physician Locator and the Naloxone Provider Guide.

INTERVENTIONS:
Behavioral: Opioid Naive, OR — Visits where the order is for an included opioid and there is no prior opioid prescription with a start date of greater than 1 day and less than 91 days and clinician is on the clinic list as a treating member of the clinic
  Arms: Behavioral Intervention Arm
Behavioral: At-risk for long-term use, OR — Visit where the order is for an included opioid, there is a prior opioid prescription with a start date greater than 1 day and less than 91 days, and there is no prior opioid prescription with a start date greater than 90 days and clinician is on the clinic list as a treating member of the clinic
  Arms: Behavioral Intervention Arm
Behavioral: Long-term opioid recipient — Total opioid doses are at least 50 MME per day, there are two or more prior opioid prescriptions with two different start dates both greater than 1 day and less than 91 days, and there is a prior opioid prescription with a start date greater than 90 days and less than 181 days and clinician is on the clinic list as a treating member of the clinic
  Arms: Behavioral Intervention Arm

SUMMARY:
The opioid epidemic has had a tremendous negative impact on the health of persons in the U.S. The objective of the trial 1 of Application of Economics & Social psychology to improve Opioid Prescribing Safety (AESOPS-T1), is to discourage unnecessary opioid prescribing through the application of "behavioral insights"-empirically-tested social and psychological interventions that affect choice.

DETAILED DESCRIPTION:
A multisite study, AESOPS-T1 randomizes clinics to behavioral intervention or control. Clinics randomized to the behavioral intervention arm receive electronic health record (EHR)-based nudges. Eligible participants are clinicians who practice ambulatory primary care at the participating clinical sites in Illinois and California. At the time of opioid prescribing, clinicians in clinics randomized to the intervention group will be prompted with an EHR nudge when the prescribing history for the patient falls into one of the following three mutually exclusive categories: Opioid naïve, At-risk for long-term use, or Long-term opioid recipient. These EHR-based nudges include accountable justification, defaults and precommitments. The control arm receives no EHR-based intervention. Both arms receive guideline education. The primary outcome is the change in clinician aggregate weekly milligram morphine equivalent (MME) dose and the secondary outcome is the proportion of dosages that equal or exceed 50 MME per day. These outcomes will be estimated by treatment arm with an intent-to-treat difference-in-differences framework using a mixed-effects regression model on clinician MME daily dose. The intervention period will be 18-months, with a 6-month follow-up period to measure the persistence of effects after the interventions conclude.

ELIGIBILITY:
Inclusion Criteria:

* Providers of clinics that see patients ≥ 18 years old and for whom clinic leadership agrees to participate.

Exclusion Criteria:

* Visits will be excluded from intervention when the patient has active cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason N Doctor, PhD, Principal Investigator — University of Southern California
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Kelley MA, Persell SD, Linder JA, Friedberg MW, Meeker D, Fox CR, Goldstein NJ, Knight TK, Zein D, Rowe TA, Sullivan MD, Doctor JN. The protocol of the Application of Economics & Social psychology to improve Opioid Prescribing Safety Trial 1 (AESOPS-1): Electronic health record nudges. Contemp Clin Trials. 2021 Apr;103:106329. doi: 10.1016/j.cct.2021.106329. Epub 2021 Feb 24. PMID 33636344
- See also: Related Info — https://doi.org/10.1016/j.cct.2021.106329

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Behavioral Intervention Arm: Clinicians in clinics randomized to the intervention group will receive guideline education and be prompted with an EHR nudge when the prescribing history for the patient falls into one of the following three categories: Opioid naïve, At-risk for long-term use, or Long-term opioid recipient.
Period: Overall Study
Arm/Group | Behavioral Intervention Arm | Control
Started | 322; 43 Clinics | 233; 43 Clinics
Completed | 275; 43 Clinics | 207; 42 Clinics
Not Completed | 47; 0 Clinics | 26; 1 Clinics
Not completed — No valid opioid prescriptions during study timeframe | 47 | 26

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Intervention Arm: Clinicians in clinics randomized to the intervention group receive guideline education and will be prompted with an EHR nudge when the prescribing history for the patient falls into one of the following three categories: Opioid naïve, At-risk for long-term use, or Long-term opioid recipient.
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention Arm | Control | Total
Number analyzed (Participants) | 322 | 233 | 555
Age, Customized [Number; unit: years]
  Unknown/Not reported | 322 | 233 | 555
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 199 | 135 | 334
  Male | 121 | 92 | 213
  Unknown/Not reported | 2 | 6 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 322 | 233 | 555

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Per-clinician Log Total Weekly MME Between Baseline and Intervention for Opioid Naïve and At-Risk Patients (Below 50 MME Daily Dose Rxs)
Description: Change = (18-month intervention average of natural log MME summed per-clinician, per-week - 6-month baseline average of natural log MME summed per-clinician, per-week). Log(total MME) = log(Rx strength x number of pills x opioid conversion factor)
Time Frame: 6-month baseline and 18-month intervention
Population: Clinicians enrolled at AltaMed and Northwestern University who prescribed an opioid Rx < 50 MME during study period. Historical Rxs, suppositories/injectionables, control clinicians who erroneously received alerts, and Rxs prescribed to patients diagnosed with cancer, or who were under 18 years, were excluded.
Measure: Mean (Standard Deviation); unit: chg in avg per-clin log total weekly MME
Arm/Group | Behavioral Intervention Arm | Control
Number analyzed (Participants) | 275 | 207
chg in avg per-clin log total weekly MME | -0.14 (0.01) | -0.05 (0.01)
Statistical Analysis 1: Comparison: Behavioral Intervention Arm vs Control; Assuming a clinic-level intraclass correlation of 0.01, alpha 0.025, 86 clinics, and 5.5 clinicians per-clinic (N = 473), it was calculated we would have over 85% power for a one-tailed test detecting a 12% reduction in MME from baseline to intervention; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Left-Censored Tobit Regression; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.12 to -0.07], Standard Error of Mean 0.01

2. Primary Outcome: Change in Average Per-clinician Log Total Weekly MME Between Baseline and Intervention for Chronic Opioid Patients (=> 50 MME Daily Dose Rxs)
Description: as for outcome 1
Time Frame: 6-month baseline and 18-month intervention
Population: Clinicians enrolled at AltaMed and Northwestern University who prescribed an opioid Rx => 50 MME during study period. Historical Rxs, suppositories/injectionables, control clinicians who erroneously received alerts, and Rxs prescribed to patients diagnosed with cancer, or who were under 18 years, were excluded.
Measure: Mean (Standard Deviation); unit: chg in avg per-clin log total weekly MME
Arm/Group | Behavioral Intervention Arm | Control
Number analyzed (Participants) | 185 | 129
chg in avg per-clin log total weekly MME | -0.21 (0.02) | -0.02 (0.01)
Statistical Analysis 1: Comparison: Behavioral Intervention Arm vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Left-Censored Tobit Regression; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.23 to -0.16], Standard Error of Mean 0.02

3. Secondary Outcome: Change in Average Per-clinician Weekly Proportion of Chronic Patients Prescribed a High Dose Opioid (=> 50 MME Daily Dose Rxs) Between Baseline and Intervention
Description: Change = (18-month intervention average per-clinician weekly proportion - 6-month baseline average per-clinician weekly proportion). Proportion = number of chronic patients who received Rx => 50 MME per-clinician, per-week/total patients who received opioid Rx per-clinician, per-week
Time Frame: 6-month baseline and 18-month intervention
Population: Clinicians enrolled at AltaMed and Northwestern University who prescribed an opioid Rx during study period. Historical Rxs, suppositories/injectionables, control clinicians who erroneously received alerts, and Rxs prescribed to patients diagnosed with cancer, or who were under 18 years, were excluded.
Measure: Mean (Standard Deviation); unit: Mean weekly proportion of chronic pts
Arm/Group | Behavioral Intervention Arm | Control
Number analyzed (Participants) | 275 | 207
Mean weekly proportion of chronic pts | -0.08 (0.01) | 0 (0.01)
Statistical Analysis 1: Comparison: Behavioral Intervention Arm vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.10 to -0.06], Standard Error of Mean 0.01

4. Other Pre Specified Outcome: Change in Average Per-clinician Log Total Weekly MME Between Baseline and Post-intervention for Opioid Naïve and At-Risk Patients (Below 50 MME Daily Dose Rxs)
Description: Change = (6-month post-intervention average of natural log MME summed per-clinician, per-week - the 18-month baseline average of natural log MME summed per-clinician, per-week). Log(total MME) = log(Rx strength x number of pills x opioid conversion factor)
Time Frame: 6-month baseline and 6-month post-intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: chg in avg per-clin log total weekly MME
Arm/Group | Behavioral Intervention Arm | Control
Number analyzed (Participants) | 275 | 207
chg in avg per-clin log total weekly MME | -0.09 (0.01) | -0.04 (0.01)
Statistical Analysis 1: Comparison: Behavioral Intervention Arm vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Left-Censored Tobit Regression; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.08 to -0.03], Standard Error of Mean 0.01

5. Other Pre Specified Outcome: Change in Average Per-clinician Weekly Proportion of Chronic Patients Prescribed a High Dose Opioid (=> 50 MME Daily Dose Rxs) Between Baseline and Post-intervention
Description: Change = (6-month post-intervention average per-clinician weekly proportion - 6-month baseline average per-clinician weekly proportion). Proportion = number of chronic patients who received Rx => 50 MME per-clinician, per-week/total patients who received opioid Rx per-clinician, per-week
Time Frame: 6-month baseline and 6-month post-intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Mean weekly proportion of chronic pts
Arm/Group | Behavioral Intervention Arm | Control
Number analyzed (Participants) | 275 | 207
Mean weekly proportion of chronic pts | -0.02 (0.01) | -0.01 (0.01)
Statistical Analysis 1: Comparison: Behavioral Intervention Arm vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.392, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to -0.01], Standard Error of Mean 0.01

6. Other Pre Specified Outcome: Change in Average Per-clinician Log Total Weekly MME Between Baseline and Post-intervention for Chronic Opioid Patients (=> 50 MME Daily Dose Rxs)
Description: Change = (6-month post-intervention average of natural log MME summed per-clinician, per-week - the 6-month baseline average of natural log MME summed per-clinician, per-week). Log(total MME) = log(Rx strength x number of pills x opioid conversion factor)
Time Frame: 6-month baseline and 6-month post-intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: chg in avg per-clin log total weekly MME
Arm/Group | Behavioral Intervention Arm | Control
Number analyzed (Participants) | 185 | 129
chg in avg per-clin log total weekly MME | -0.13 (0.01) | -0.04 (0.02)
Statistical Analysis 1: Comparison: Behavioral Intervention Arm vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Left-Censored Tobit Regression; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.13 to -0.05], Standard Error of Mean 0.02

ADVERSE EVENTS:
Time Frame: 18 month intervention period
Arm/Group | Behavioral Intervention Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/322 | 0/233
Serious Adverse Events (participants affected / at risk) | 0/322 | 0/233
Other Adverse Events (participants affected / at risk) | 0/322 | 0/233

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT04477304/Prot_SAP_000.pdf